CLINICAL TRIAL: NCT00002359
Title: A Multicenter, Double-Blind, Phase III, Adjuvant-Controlled Study of the Effect of 10 Units of HIV-1 Immunogen (Remune) Compared to Incomplete Freund's Adjuvant (IFA) Alone Every 12 Weeks on AIDS-Free Survival in Subjects With HIV Infection and CD4 T-Lymphocytes Between 300 and 549 Cells/microL Regardless of Concomitant HIV Therapies
Brief Title: A Multicenter, Double-Blind, Phase III, Adjuvant-Controlled Study of the Effect of 10 Units of HIV-1 Immunogen (Remune) Compared to Incomplete Freund's Adjuvant (IFA) Alone Every 12 Weeks on AIDS-Free Survival in Subjects With HIV Infection and CD4 T-Lymphocytes Between 300 and 549 Cells/microL Rega
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Immune Response Corporation (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 092; 806
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-06

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Viral Vaccines; HIV-1; AIDS-Related Complex; AIDS Vaccines; Salk HIV Immunogen
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — HIV-1 immunogen, incomplete Freund's adjuvant

INTERVENTIONS:
Biological: HIV-1 Immunogen

SUMMARY:
To determine the effect of HIV-1 immunogen (Remune) on AIDS-free survival, defined as the time prior to development of an AIDS-defining condition or death.

DETAILED DESCRIPTION:
Patients receive 10 units of HIV-1 immunogen in IFA or IFA alone every 12 weeks, then are followed for 104-148 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretrovirals if on a stable dose for at least the past 3 months.

Patients must have:

* HIV-1 infection with CD4 count 300-549 cells/mm3.
* No AIDS-defining condition.
* Been on a stable dose of antiretroviral for the past 3 months, if taking antiretrovirals.

NOTE:

* KS is permitted if not requiring systemic therapy.

Prior Medication:

Allowed:

* Prior antiretrovirals.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Systemic chemotherapy for KS.
* Treatment for malignancy other than basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.

Patients with the following prior conditions are excluded:

* History of any illness that would interfere with study.
* Acute infection requiring prescription therapy within the past month, other than genital herpes and oral or vaginal candidiasis.

Prior Medication:

Excluded:

* Prior HIV-1 Immunogen. Unwilling to use effective safe sex practices. Active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000

CONTACTS AND LOCATIONS:
Locations (54):
- United States (54):
  - Phoenix Body Positive, Phoenix, Arizona
  - Ctr for Special Immunology, Irvine, California
  - Jeffrey Goodman Special Care Clinic, Los Angeles, California
  - Kraus Med Partners, Los Angeles, California
  - Cedars Sinai Med Ctr, Los Angeles, California
  - AIDS Community Research Consortium, Redwood City, California
  - Whitman Walker Clinic Inc, Washington D.C., District of Columbia
  - Anderson Clinical Research, Washington D.C., District of Columbia
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Ctr for Special Immunology, Miami Beach, Florida
  - The Coleman Institute, North Miami, Florida
  - Clinical Pharmacology Services, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Rush Med Ctr, Chicago, Illinois
  - Chicago AIDS Research Alliance, Chicago, Illinois
  - Ctr for Special Immunology, Chicago, Illinois
  - Community Hosp Indianapolis, Indianapolis, Indiana
  - UKSM-W Med Practice Association, Wichita, Kansas
  - Univ of Kentucky / Division of ID Research, Lexington, Kentucky
  - JSI Research and Training Institute, Boston, Massachusetts
  - Community Research Initiative of New England, Brookline Village, Massachusetts
  - Providence Mercy Hosp, Holyoke, Massachusetts
  - Wayne State Univ / WSU / DMC HIV / AIDS Program, Detroit, Michigan
  - Henry Ford Hosp / Infectious Diseases, Detroit, Michigan
  - Abbott Northwestern Hosp, Minneapolis, Minnesota
  - Kansas City AIDS Research Consortium, Kansas City, Missouri
  - Washington Univ / St Louis Connect Care, St Louis, Missouri
  - Anderson Clinical Research, New York, New York
  - St Luke's - Roosevelt Hosp Ctr / Div of Infect Dis, New York, New York
  - Cornell Univ Med College, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Dr Barbara Justice, New York, New York
  - Community Health Network, Rochester, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Nalle Clinic, Charlotte, North Carolina
  - Univ of Cincinnati Med Ctr / Holmes Division, Cincinnati, Ohio
  - Ohio State Univ / Division of Infectious Disease, Columbus, Ohio
  - Univ of Oklahoma, Oklahoma City, Oklahoma
  - The Research and Education Group, Portland, Oregon
  - The Graduate Hosp, Philadelphia, Pennsylvania
  - Anderson Clinical Research, Pittsburgh, Pennsylvania
  - Mem Hosp of Rhode Island, Pawtucket, Rhode Island
  - Med Univ of South Carolina, Charleston, South Carolina
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Metroplex Clinical Research Ctr, Dallas, Texas
  - Univ of Texas Med Branch Ctr for Clinical Studies, Galveston, Texas
  - ONCOL Med Associates / PA, Houston, Texas
  - Univ of Utah Med School / Clinical Trials Ctr, Salt Lake City, Utah
  - Infectious Disease Physicians Inc, Annandale, Virginia
  - Hampton Roads Med Specialists, Hampton, Virginia
  - Eastern Virginia Med School, Norfolk, Virginia
  - Novum Inc, Seattle, Washington
  - Wisconsin AIDS Research Consortium, Milwaukee, Wisconsin

REFERENCES:
- [Background] Kahn JO, Cherng DW, Mayer K, Murray H, Lagakos S. Evaluation of HIV-1 immunogen, an immunologic modifier, administered to patients infected with HIV having 300 to 549 x 10(6)/L CD4 cell counts: A randomized controlled trial. JAMA. 2000 Nov 1;284(17):2193-202. doi: 10.1001/jama.284.17.2193. PMID 11056590
- [Derived] Rao MP, Al-Khatib SM, Pokorney SD, She L, Romanov A, Nicolau JC, Lee KL, Carson P, Selzman CH, Stepinska J, Cleland JG, Tungsubutra W, Desvigne-Nickens PM, Sueta CA, Siepe M, Lang I, Feldman AM, Yii M, Rouleau JL, Velazquez EJ; STICH Trial Investigators. Sudden Cardiac Death in Patients With Ischemic Heart Failure Undergoing Coronary Artery Bypass Grafting: Results From the STICH Randomized Clinical Trial (Surgical Treatment for Ischemic Heart Failure). Circulation. 2017 Mar 21;135(12):1136-1144. doi: 10.1161/CIRCULATIONAHA.116.026075. Epub 2017 Feb 2. PMID 28154006